CLINICAL TRIAL: NCT05880264
Title: Development of Standard References of Maximal Inspiratory Pressure and Maximal Expiratory Pressure in Healthy Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0745
Record Dates: First submitted 2023-03-26; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
(1) Maximum respiratory pressure (MRP)1) Maximum inspiratory pressure (maximum intake pressure) and maximum expiratory pressure (MEP) Digital spirometer (Pony FX, COSMED Inc., Italy) are used to measure the micro-paste in a seated position. MIP is based on the pressure maintained for at least 1 second, inhaling or exhaling with maximum effort in the maximum exhalation state (=residual volume) and the maximum exhalation state (=total lung capacity). The maximum positive pressure value of the MEP and the minimum sound pressure value of the MIP are selected among the three or more attempts. 2) Using the MVV (maximum volitional ventilation) Digital spirometer (Pony FX, COSMED Inc., Italy) machine, repeat breathing deeply and quickly for 12 seconds while wearing a nose plug, and multiply it by 5 to obtain the L/min value. (2) Measure the values of the Pneumatic ventilation. · FVC (forced vital capacity): Total expiratory volume of one of the maximum effort gases · FEV1 (forced expiratory volume 1, effort expiratory volume): Ejected expiratory volume of the first second of the maximum effort expiratory volume (FEV1/FVC): FVC ratio, percentage of FVCs, and extraction of the FVC (excessive flow). PEF): Highest speed of effort opportunity

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 65 years old.
2. a patient under general anesthesia
3. Patients in ASA class I to II
4. a patient with no history of thoracic anatomy or surgery
5. Patients with normal chest X-ray findings for preoperative evaluation.

Exclusion Criteria:

1. Patients with no natural history of thoracic abnormalities or surgery
2. Patients with asthma, pneumonia, tuberculosis, pneumothorax, chronic obstructive pulmonary disease and epileptic pulmonary disease
3. Patients who have difficulty communicating with the examiner.

Ages: 19 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who are scheduled to surgery under general anesthesia at Yonsei University Severance Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Measure MIP for healthy Koreans and obtain the reference value | up to 1 year
  A. The subject sits on a chair and covers his nose with a nose plug. B. The patient prepares the test with the Pony Fx MIP/MEP spirometer connected filter in his mouth.
  C. After inhaling as much as possible, exhale strongly through the filter with maximum force.
  D. At this time, the assistant guides the patient from the side so that the patient can exhale with maximum force.
  E. Check the results and select a pressure that is maintained for at least 1 second.
  F. The minimum sound pressure value is selected by attempting the A~E process more than three times.
Measure MEP for healthy Koreans and obtain the reference value. | up to 1 year
  A. The subject sits on a chair and covers his nose with a nose plug. B. The patient prepares the test with the Pony Fx MIP/MEP spirometer connected filter in his mouth.
  C. Breathe out as much as you can, and then breathe in strongly through the filter with maximum force.
  D. At this time, the assistant guides the patient from the side to breathe in with maximum force.
  E. Check the results and select a pressure that is maintained for at least 1 second.
  F. The maximum positive pressure value is selected by trying the A~E process more than three times.
Measure MVV for healthy Koreans and obtain the reference value. | up to 1 year
  A. The subject sits on a chair and covers his nose with a nose plug. B. The patient prepares the test with the Pony Fx MIP/MEP spirometer connected filter in his mouth.
  C. Repeat deep and fast breathing for 12 seconds with the start of the test. D. At this time, the assistant looks at the result graph and guides the patient from the side to make the best effort until the end.
  E. Multiply the result for 12 seconds by 5 to obtain the L/min value of MVV.

SECONDARY OUTCOMES:
Check the predictive equation (forced vital capacity) | up to 1 year
  Measure the above values using a Pulmonary function test Digital spirometer (Pony FX, COSMED Inc., Italy) machine.
  * FVC (forced vital capacity): Total expiratory volume of one of the maximum effort gases
  * FEV1 (forced expiratory volume 1, effort expiratory volume): Ejected expiratory volume of the first second of the maximum effort expiratory volume (FEV1/FVC): FVC ratio, percentage of FVCs, and extraction of the FVC (excessive flow).
  PEF): Highest speed of effort opportunity
Check the predictive equation (forced expiratory volume 1) | up to 1 year
  Measure the above values using a Pulmonary function test Digital spirometer (Pony FX, COSMED Inc., Italy) machine.
  * FVC (forced vital capacity): Total expiratory volume of one of the maximum effort gases
  * FEV1 (forced expiratory volume 1, effort expiratory volume): Ejected expiratory volume of the first second of the maximum effort expiratory volume (FEV1/FVC): FVC ratio, percentage of FVCs, and extraction of the FVC (excessive flow).
  PEF): Highest speed of effort opportunity
Check the predictive equation (FEV1/FVC) | up to 1 year
  Measure the above values using a Pulmonary function test Digital spirometer (Pony FX, COSMED Inc., Italy) machine.
  * FVC (forced vital capacity): Total expiratory volume of one of the maximum effort gases
  * FEV1 (forced expiratory volume 1, effort expiratory volume): Ejected expiratory volume of the first second of the maximum effort expiratory volume (FEV1/FVC): FVC ratio, percentage of FVCs, and extraction of the FVC (excessive flow).
  PEF): Highest speed of effort opportunity
Check the predictive equation (PEF) | up to 1 year
  Measure the above values using a Pulmonary function test Digital spirometer (Pony FX, COSMED Inc., Italy) machine.
  * FVC (forced vital capacity): Total expiratory volume of one of the maximum effort gases
  * FEV1 (forced expiratory volume 1, effort expiratory volume): Ejected expiratory volume of the first second of the maximum effort expiratory volume (FEV1/FVC): FVC ratio, percentage of FVCs, and extraction of the FVC (excessive flow).
  PEF): Highest speed of effort opportunity

CONTACTS AND LOCATIONS:
Overall Officials: HYO JIN BYON, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No